CLINICAL TRIAL: NCT07206277
Title: Use of Transient Elastography to Guide Immunosuppression Minimization Post Liver Transplantation
Brief Title: Fibroscan to Guide Post Transplant Immunosuppression Minimization
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00148986
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Immunosuppression
Keywords: Liver transplantation; minimization; rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Followed per standard of care
- Immunosuppression minimization (Experimental): will have immunosuppression reduction during the study using fibroscan
  Interventions: Other: Immunosuppression reduction

INTERVENTIONS:
Other: Immunosuppression reduction — In patients with LSM < 8.4 kPa we will gradually reduce IS by 30% (e.g. if on tacrolimus 6 mg daily, dose will be reduced to 4 mg daily) over three months. In patients with immunosuppression reduction we will perform TE at 4, 7 and 12 months after IS reduction to ensure there is no change in LSM. We will get liver biochemistry every 2 weeks x 4 months to ensure labs remain within normal range. Following this, patients will resume monthly labs.
  Arms: Immunosuppression minimization

SUMMARY:
Following Liver transplantation, recipients remain on life long immunosuppression. Prolonged exposure to immunosuppression is associated with side effects and complications including kidney dysfunction, diabetes, heart disease and cancer risk.

Therefore studies are looking at safe ways to reduce or stop immunosuppression. An individual without autoimmune liver disease (these patients are at higher risk of rejection), without history of rejection, with normal blood tests (liver biochemistry, liver function, etc.) can be eligible for minimization of immunosuppression. A recent study showed use of fibroscan (an Ultrasound, which provides information on liver stiffness (diseased liver is hard while a normal liver is soft) and fat content) provides more objective information to help investigators select individuals who will tolerate immunosuppression minimization.

Our goal is to see if use of fibroscan allows the investigators to safely minimize immunosuppression in eligible individuals. The secondary aims are to assess benefit on kidney function, heart disease and risk factors for heart disease.

DETAILED DESCRIPTION:
Excellent short-term survival following liver transplantation (LT) has translated into long-term survival with many patients surviving over 25 years (1). Thus, many patients will have prolonged exposure to immunosuppression (IS), which is a double edged sword and needs to be carefully balanced; inadequate levels may lead to rejection whereas consistently high levels may lead to side effects and long term complications (e.g. metabolic syndrome (MS), renal dysfunction (CKD), cardiovascular disease (CVD), malignancy) (2). Of note, the type of IS used (mTOR inhibitors (mTOR) vs. calcineurin inhibitors (CNI)) may also contribute to complications. Whereas CNI use is associated with renal dysfunction and development of de novo steatosis (3), mTOR use is associated with increased risk of dyslipidemia; combined use of CNI and mTOR has been shown to lead to hyperglycemia (4, 5). Not surprisingly, IS use is associated with development of MS post LT (2, 6). Due to shared risk factors, presence of steatosis may also lead to increased risk of MS, CVD and renal dysfunction. Thus, minimization of IS may lead to reduced complications. Management of IS varies by transplant centre and involves trial and error; most rely on drug levels, liver biochemistry, indication for transplant, duration following transplant, and demographics of the recipient. Changes in IS tend to be reactive in nature and occur in the setting of complications. Studies have shown a substantial number of patients may be able to tolerate lower levels of IS (7, 8). Thus, there is a need for an objective, non-invasive, measure that can help clinicians optimize IS.

Vibration-Controlled Transient elastography (TE; FibroScan®) is a promising tool; it is a non-invasive technique for assessment of liver stiffness measurement (LSM) that additionally provides the controlled attenuation parameter (CAP), which reflects hepatic steatosis. TE accurately predicts degree of liver fibrosis and portal hypertension regardless of etiology of liver disease (9-11). In the pre-transplant setting it is a common point-of-care tool that has led to reduced need for liver biopsy, risk stratification of patients with non-alcoholic fatty liver disease (12), and use as a guide to treat patients with Hepatitis B infection (13).

The use of TE post LT remains limited with a scarcity of studies. The few studies that exist are limited by a small sample size and short follow up post-LT. Nevertheless, these studies show there is a correlation between TE and severity of acute cellular rejection (r=0.6; p< 0.001) (10); fibrosis and degree of portal hypertension (14); association with other diseases (idiopathic hepatitis, steatohepatitis, cholangitis, de novo or recurrent disease) (9); association with steatosis (AUROC 0.88) (15); and association with decompensation and graft/patient survival (16).

In a recent study, TE was used to identify individuals with low risk of rejection who could safely undergo IS minimization. Authors showed that subclinical allo-immune injury was associated with increased LSM and that patients with LSM below 8.4 kPa had a negligible probability of having active alloimmune damage (11%); these patients could potentially have reduction of IS (7). This study provides the scientific basis for assessing the use of TE as a guide to IS management.

The aim of this study is to assess if TE can be used to safely guide IS minimization in stable post-LT patients. The secondary aims will include impact on renal function, MS, CVD, malignancy, graft and patient survival. In a nested study, the investigators will explore the use of TE to investigate the effect of type of immunosuppression used and the development of hepatic steatosis, based on the CAP score (nested case-control study).

ELIGIBILITY:
Inclusion Criteria:

* 2 years or more post-liver transplant
* 18 years or older

Exclusion Criteria:

* diagnosis of either acute or chronic rejection in the past 12 months
* abnormal liver enzymes (ALT > 50; bilirubin > 19 umol/L)
* transplant for autoimmune liver disease (autoimmune hepatitis, primary sclerosing cholangitis, and primary biliary cholangitis)
* presence of HCV RNA
* presence of HBV DNA
* presence of class II donor specific antibodies (DSA; pre-existing or de novo)
* beyond 6 years of transplantation
* presence of ascites, decompensated heart failure, biliary obstruction, CKD (bl eGFR 30 ml/min/1.73m2 or less), re-transplantation, or multi-visceral transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants successfully achieving immunosuppression minimization | Immunosuppression reduced over 3 months. Follow up to ensure no rejection at 6 months.
  Goal 30% reduction in immunosuppression without rejection

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided